CLINICAL TRIAL: NCT02442661
Title: Clinical Validation of a Predictive Model for the Presence of Cervical Lymph Node Metastasis in Papillary Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-2053
Record Dates: First submitted 2015-04-22; First posted 2015-05-13 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research study is performed to compare the accuracy of two methods of lymph node evaluation: research method versus standard method. Standard method is what is usually performed as standard of care where the radiologist evaluates the images overall and decides whether each node seen should or should not be biopsied. In the research method, a second radiologist will evaluate the ultrasound images of the lymph nodes separately, and use a small specific checklist of ultrasound appearance to determine whether each node should or should not be biopsied. Results of both the standard and research method will be used to decide which node(s), if any should be biopsied. Neck ultrasound examination, lymph node evaluation by standard method and subsequent lymph node biopsy are part of the standard clinical care. It is less likely but possible that the research method may identify additional lymph nodes for biopsy to check if that lymph node contains thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTC and at least one sonographic examination of the cervical lymph nodes.
* Patients can only be included in the study once. Thus, if they have two sonographic examinations, only one can be included in the study results.
* All patients who fit the study criteria after the start of the study will be included, using the first sonographic exam as the study exam.

Exclusion Criteria:

* Lymph node with oval shape, hypoechoic cortex, smooth border, hyperechoic hilum and hilar Doppler flow by ultrasound are considered to be normal and be excluded from FNAB per standard clinical practice.
* Lymph node less than 5 mm in short axis on ultrasound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-thyroidectomy patients with a pathological diagnosis of Papillary Thyroid Cancer (PTC) who undergo cervical lymph node evaluation for detection of locoregional metastasis will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Detection of lymph node metastasis in a patient with Papillary Thyroid Cancer by neck ultrasound by radiologist's standard assessment method (Ir test). | 6 months
Detection of lymph node metastasis in a patient with Papillary Thyroid Cancer by neck ultrasound by predictive model method (Im test). | 6 months

SECONDARY OUTCOMES:
Confirmation of the lymph node metastasis by fine needle aspiration biopsy prior to the surgery. | 6 months
Measure true positive and false positive results of Ir test and Im test for comparison. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nayana Patel, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Rebecca J Guigli, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Participant data is only available to study personnel